CLINICAL TRIAL: NCT01273246
Title: A Blind, Randomized and Placebo-controlled Clinical Trial With Inactivated Enterovirus Type 71 Vaccines in Healthy Children.
Brief Title: Safety of an Inactivated Enterovirus Type 71 Vaccines in Healthy Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EV71-1001-Ib
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2011-07

CONDITIONS: Hand-foot-mouth Disease; Infection; Viral, Enterovirus
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Infections; Enterovirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Children Group 1: 200U EV71 vaccine (Experimental): 12 children received 3 doses of 200U EV71 vaccine 28 days apart
  Interventions: Biological: 200U inactivated Enterovirus Type 71 Vaccine
- Children Group 1: Placebo (Placebo Comparator): 6 children received 3 doses of placebo 28 days apart
  Interventions: Biological: Placebo
- Children Group 2: 400U EV71 vaccine (Experimental): 12 children received 3 doses of 400U EV71 vaccine 28 days apart
  Interventions: Biological: 400U inactivated Enterovirus Type 71 Vaccine
- Children Group 2: Placebo (Placebo Comparator): 6 children received 3 doses of placebo 28 days apart
  Interventions: Biological: Placebo
- Infants Group 1: 100U EV71 vaccine (Experimental): 24 infants received 3 doses of 100U EV71 vaccine 28 days apart
  Interventions: Biological: 100U inactivated Enterovirus Type 71 Vaccine
- Infants Group 1: Placebo (Placebo Comparator): 8 infants received 3 doses of placebo 28 days apart
  Interventions: Biological: Placebo
- Infants Group 2: 200U EV71 vaccine (Experimental): 24 infants received 3 doses of 200U EV71 vaccine 28 days apart
  Interventions: Biological: 200U inactivated Enterovirus Type 71 Vaccine
- Infants Group 2: Placebo (Placebo Comparator): 8 infants received 3 doses of placebo 28 days apart
  Interventions: Biological: Placebo
- Infants Group 3: 400U EV71 vaccine (Experimental): 24 infants received 3 doses of 400U EV71 vaccine 28 days apart
  Interventions: Biological: 400U inactivated Enterovirus Type 71 Vaccine
- Infants Group 3: Placebo (Placebo Comparator): 8 infants received 3 doses of placebo 28 days apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 100U inactivated Enterovirus Type 71 Vaccine — Inactivated Enterovirus Type 71 Vaccine, 100U per 0.5ml per dose. Vaccine will be administered as a single 0.5 mL intramuscular injection in the deltoid muscle of the arm
  Other Names: EV71 vaccine
  Arms: Infants Group 1: 100U EV71 vaccine
Biological: 200U inactivated Enterovirus Type 71 Vaccine — Inactivated Enterovirus Type 71 Vaccine, 200U per 0.5ml per dose. Vaccine will be administered as a single 0.5 mL intramuscular injection in the deltoid muscle of the arm
  Other Names: EV71 vaccine
  Arms: Children Group 1: 200U EV71 vaccine; Infants Group 2: 200U EV71 vaccine
Biological: 400U inactivated Enterovirus Type 71 Vaccine — Inactivated Enterovirus Type 71 Vaccine, 400U per 0.5ml per dose. Vaccine will be administered as a single 0.5 mL intramuscular injection in the deltoid muscle of the arm
  Other Names: EV71 vaccine
  Arms: Children Group 2: 400U EV71 vaccine; Infants Group 3: 400U EV71 vaccine
Biological: Placebo — Placebo, all components of the trial vacccine except for the Enterovirus Type 71 virus antigen, 0.5ml per dose. Placebo will be administered as a single 0.5 mL intramuscular injection in the deltoid muscle of the arm
  Arms: Children Group 1: Placebo; Children Group 2: Placebo; Infants Group 1: Placebo; Infants Group 2: Placebo; Infants Group 3: Placebo

SUMMARY:
A Phase I clinical trialto evaluate the safety of an Inactivated Enterovirus Type 71 Vaccine in healthy children (3-11y) and infants (6-35m).

DETAILED DESCRIPTION:
36 eligible children aged from 3 to 11 years and 96 eligible infants aged from 6 to 35 months will be enrolled in the study, they will be randomized to receive different dosage of vaccine candidate or placebo to evaluate the safety of this vaccine

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, aged from 6 months to 11 years old Health is determined by medical history, physical examination, laboratory examination and clinical judgment of the investigator
2. Provided legal identification for the sake of recruitment.
3. Subjects and/or parent(s)/legal guardian(s) are able to understand and sign informed consents.
4. Birth weight more than 2500 grams

Exclusion Criteria:

1. Histroy of Hand-foot-mouth Disease
2. Subject that has allergic history of vaccine, or allergic to any ingredient of vaccine
3. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
4. Congenital malformations or developmental disorders, genetic defects, or severe malnutrition
5. Epilepsy, seizures or convulsions history, or family history of mental illness
6. Autoimmune disease or immunodeficiency, or parents, brothers and sisters have autoimmune diseases or immunodeficiency
7. History of asthma, angioedema, diabetes or malignancy
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
10. Asplenia, functional asplenia or any condition resulting in the absence or removal the spleen
11. Acute illness or acute exacerbation of chronic disease within the past 7 days
12. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
13. History of any blood products within 3 months
14. Administration of any live attenuated vaccine within 28 days
15. Administration of subunit or inactivated vaccines ,e.g., pneumococcal vaccine, or allergy treatment within 14 days
16. Axillary temperature > 37.0 centigrade before vaccination
17. Abnormal laboratory parameters before vaccination
18. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the inactivated Enterovirus Type 71 Vaccine | 6 months
  All adverse events were records. Blood cell and biochemistry were performed.

SECONDARY OUTCOMES:
To evaluate the immunogenicity of the inactivated Enterovirus Type 71 Vaccine | 6 months
  virus neutralization assays were performed.

CONTACTS AND LOCATIONS:
Overall Officials: Yan-pin Li, MD, Principal Investigator — Guangxi Centers for Disease Control and Prevention
Locations (1):
- GuangXi Center for Diseases Control and Prevention, Nanning, Guangxi, China

REFERENCES:
- [Derived] Mao Q, Cheng T, Zhu F, Li J, Wang Y, Li Y, Gao F, Yang L, Yao X, Shao J, Xia N, Liang Z, Wang J. The cross-neutralizing activity of enterovirus 71 subgenotype c4 vaccines in healthy chinese infants and children. PLoS One. 2013 Nov 19;8(11):e79599. doi: 10.1371/journal.pone.0079599. eCollection 2013. PMID 24260259
- [Derived] Li YP, Liang ZL, Gao Q, Huang LR, Mao QY, Wen SQ, Liu Y, Yin WD, Li RC, Wang JZ. Safety and immunogenicity of a novel human Enterovirus 71 (EV71) vaccine: a randomized, placebo-controlled, double-blind, Phase I clinical trial. Vaccine. 2012 May 9;30(22):3295-303. doi: 10.1016/j.vaccine.2012.03.010. Epub 2012 Mar 15. PMID 22426327